CLINICAL TRIAL: NCT04287413
Title: Determining the Impact of a New Physiotherapist-led Primary Care Model for Low Back Pain - a Cluster Randomized Controlled Trial
Brief Title: Determining the Impact of a New Physiotherapist-led Primary Care Model for Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan Miller, PT, PhD (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Jordan Miller, PT, PhD, Assistant Professor, School of Rehabilitation Therapy, Queen's University, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REH-755-19
Record Dates: First submitted 2020-01-14; First posted 2020-02-27 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Back Pain, Low
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized controlled trial randomizing 20 sites to the PT-led primary care model for back pain or to the usual care model
Masking Description: Due to the nature of the new model of care and comparison, it is not possible to blind the patients or health care providers. Since the primary outcomes are self-reported outcome measures, the assessor is also not blind to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physiotherapist-led primary care model for back pain (Experimental): The index intervention will incorporate a PT within the primary care team and make them available at the first point of contact for people with low back pain. There will be 4 key components of this intervention: 1) Initial assessment and screening; 2) Brief individualized intervention at first visit; 3) Health services navigation; 4) Providing additional PT care for people with an unmet need (e.g., no insurance coverage for PT).
  Interventions: Behavioral: Physiotherapist-led primary care model for back pain
- Usual care (Active Comparator): The physician-led primary care intervention will be unstandardized to best reflect standard clinical practice in Canada. This usually includes a visit to a primary care physician, who would perform a history and physical examination, provide LBP education, order diagnostic imaging, prescribe medications and/or refer based on their assessment findings and patient preferences.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Physiotherapist-led primary care model for back pain — Assessment and screening: taking a history; screening for red flags, comorbidities, and risk factors of ongoing pain and disability; physical examination.
  Brief individualized intervention at the first visit: effective communication, cognitive reassurance, a few exercises, and advice/strategies to stay active.
  Health services navigation: PT assistance with navigating healthcare services based on the assessment findings. First, red-flags requiring emergency or urgent referrals. Next, comorbid conditions that would benefit from care from other healthcare providers. Finally, referral to PT (if appropriate).
  Providing additional physiotherapy care to people with an unmet need: Additional physiotherapy care will be provided to patients who have an identified need for physiotherapy but no physiotherapy coverage through private or government health insurance plans.
  Arms: Physiotherapist-led primary care model for back pain
Behavioral: Usual care — The physician led primary care intervention will be unstandardized to best reflect standard clinical practice in Canada.
  Arms: Usual care

SUMMARY:
This is a cluster randomized controlled trial to to evaluate the individual and health system impacts of implementing a new physiotherapist-led primary care model for back pain in Canada.

DETAILED DESCRIPTION:
This study aims to evaluate the individual health outcomes and health system impacts of implementing a new physiotherapist-led primary care model for people with low back pain (LBP).

The overarching goal of this study is to determine the impact of integrating a physiotherapist (PT) within primary care teams for people with LBP and making them available to patients as the first point of contact. The specific aims of the research are to determine:

1. Whether a PT-led primary care model for LBP is effective at improving function (primary outcome), pain intensity, quality of life, global rating of change, and adverse events in comparison to usual physician led primary care.
2. The impact of a PT led primary care model for LBP on the healthcare system and society (healthcare access, primary care physician workload, healthcare utilization, missed work, and cost-effectiveness). A process evaluation will assess the healthcare delivered, potential mechanisms, context of implementation, and perspectives of patients and primary care providers towards the PT-led primary care model.

ELIGIBILITY:
Inclusion Criteria:

* Adults (19 years and over) with low back pain of any duration who are seeking primary care for back pain at a participating site (primary care visit may be a first or repeat visit).

Exclusion Criteria:

* Patients who do not consent to participation
* Patients who report being unable to understand, read, and write English
* Patients for whom the cause of their back pain is cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1560 (Estimated)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Self-reported Disability | Change from baseline at 6-week, 12-week, 6-month, 9-month, and 12-month follow-ups
  Measured using the Roland Morris Disability Questionnaire (0 to 24 with higher scores indicating greater disability)
Self-reported Pain Intensity | Change from baseline at 6-week, 12-week, 6-month, 9-month, and 12-month follow-ups
  Measured using a numeric pain rating scale from 0 to 10 with higher scores indicating greater pain intensity (measured at rest, during walking, and during a lifting task)
Health Related Quality of Life | Change from baseline at 6-week, 12-week, 6-month, 9-month, and 12-month follow-ups
  Measured using the EuroQoL-5D-5L (0 to 100 with greater scores indicating greater self-reported health related quality of life)
Pain Self Efficacy | Change from baseline at 6-week, 12-week, 6-month, 9-month, and 12-month follow-ups
  Confidence in abilities to participate in usual activities using the Pain Self Efficacy Questionnaire (0-60 score with higher scores indicating higher level of confidence in dealing with pain)
Global Rating of Change | Change from baseline at 6-week, 12-week, 6-month, 9-month, and 12-month follow-ups
  Measured using an 11-point scale (-5 to +5 with negative scores indicating a worsening of physical functioning related to back pain and positive scores indicating an improvement of physical functioning related to back pain)
Satisfaction with Health Care | 6-week, 12-week, 6-month, 9-month, and 12-month follow-ups
  Measured using an 11-point scale(-5 to +5 with negative scores indicating a dissatisfaction with health care received and positive scores indicating satisfaction with health care received)
Fear of Movement | Change from baseline at 6-week, 12-week, 6-month, 9-month, and 12-month follow-ups
  Measured using the Tampa Scale of Kinesiophobia (TSK-11) [an 11-item questionnaire]. Score of 11-44 with lower scores indicating less pain-related fear. The initial protocol indicated our intention to use the TSK-17, but we changed to the TSK-11 to reduce response burden prior to initiating patient recruitment.
Catastrophic Thinking | Change from baseline at 6-week, 12-week, 6-month, 9-month, and 12-month follow-ups
  Measured using the Pain Catastrophizing Scale (0 to 52 with higher scores indicating greater catastrophic thinking)
Depressive Symptoms | Change from baseline at 6-week, 12-week, 6-month, 9-month, and 12-month follow-ups
  Measured using the 2-item Patient Health Questionnaire (PHQ-2) (0 to 6 with greater scores indicating increased depressive symptoms). This measure was changed from the PHQ-9 to PHQ-2 after initial trial registration but prior to initiating patient recruitment reduce response burden.
Adverse Events | 6-week, 12-week, 6-month, 9-month, and 12-month follow-ups
  Measured using an adverse events questionnaire that asks 1) if the patient has experienced any adverse events as a result of the treatments received (yes/no); 2) how long the event lasted (hours or days); 3) how severe the adverse event was (0-10 scale); 4) what adverse events were experienced.

SECONDARY OUTCOMES:
Health Care Accessibility | Baseline
  Percentage of patients receiving care within 48 hours.
Access to Physiotherapy Services | Baseline
  Percentage of patients who score medium or high risk on the STarT Back tool who receive physiotherapy care.
Health care utilization - electronic medical record (EMR) | 12 months
  Measuring health care utilization, from the participant's EMR, of consultations with primary care team members and access to programs offered within primary care
Health care utilization - self report | 12 months
  Measuring health care utilization (self-report survey): visits to health professionals outside of the primary care team (e.g. chiropractors, massage therapists, occupational therapists, physiotherapists, social workers), medication use, and visits to walk-in clinics.
Health care utilization - self-report | 12 months
  Measuring health care utilization from self-report survey: diagnostic imaging for the spine, pain injections or interventional procedures received, specialist visits for low back pain, hospital stays related to back pain and dysfunction, and emergency department visits for back pain. The collection of this healthcare utilization data changed from using health administrative data in Ontario accessed through the Institute for Clinical Evaluative Sience (IC/ES) to using a self-report survey prior to the initiation of patient recrutiment when we recruited sites in British Columbia.
Costs | 12 months
  Includes all health care costs (including: primary care visits, emergency department visits, hospitalizations, surgeries, consultations with other health care providers, diagnostic imaging, medications, and other care received by the patient) plus societal costs using a human capital approach for loss of productivity.
Medications Prescribed for Back Pain | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-ups
  Measured as a process outcome - medications prescribed for back pain will be collected in table format from the EMR.
Number of Diagnostic Imaging Tests Ordered | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Measured as a process outcome - the number of diagnostic imaging tests ordered will be collected in table format from the EMR.
Number of Referrals Made to Other Health Care Providers | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Measured as a process outcome - the number of referrals made to other health care providers will be collected in table format from the EMR.
Number of Notes Written to Employers or Insurers | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Measured as a process outcome - the number of notes written to employers or insurers will be collected in table format from the EMR.
Education Provided by Health Care Provider | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Measured as a process outcome (yes or no) and collected in table format from from the EMR
Exercises Prescribed | Baseline, 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Measured as a process outcome and collected in table format from the EMR
Self-Report Time Lost | 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Self-reported time lost from work, volunteering, homemaking, and educational activities
Self-Report Assistance Needed for Activities of Daily Living | 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Self-reported assistance needed, due to LBP, for self-care, housework, shopping, or transportation. Participants indicates on survey what they needed assistance for.
Extra Expenses | 6-week, 12-week, 6-month, 9-month, and 12-month follow-up
  Any extra expenses incurred as a result of LBP. Self-report

OTHER OUTCOMES:
Comorbidities | Baseline
  Measured at baseline using the Functional Comorbidity Index (an 18-item list of comorbidities that are associated with physical functioning).
Baseline characteristics | Baseline
  To describe the study population, the investigators will capture the following through the survey: age, sex, gender, identification as indigenous (First Nations, Inuit, Métis), duration and history of LBP, level of education achieved, household income, and work status.
Risk of persistent pain and disability | Baseline
  Measured using the STaRT Back tool to group participants into low, medium, and high risk groups
Participant Treatment Fidelity | 6-weeks
  Self-report adherence to physiotherapy advice

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Miller, PhD, Principal Investigator — Queen's University
Locations (2):
- Canada (2):
  - Interior Health, Kelowna, British Columbia
  - Queen's University, Kingston, Ontario

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data with other researchers.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT04287413/Prot_SAP_000.pdf